CLINICAL TRIAL: NCT04991597
Title: The Effects of Injection Site Cooling and Solution Buffering on Perceived Pain During Local Anesthesia Administration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Shift in research focus
Sponsor: Nicholas Bastidas (Other)
Responsible Party: Sponsor-Investigator, Nicholas Bastidas, Associate Professor of Plastic Surgery, Northwell Health
Organization: Northwell Health (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: LESB 001
Record Dates: First submitted 2021-08-03; First posted 2021-08-05 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Pain
Keywords: Local Anesthesia; Lidocaine; Bicarbonate; Pain; Buffering; Injection Site Cooling
MeSH Terms: conditions — Pain | interventions — Sodium Bicarbonate

STUDY DESIGN:
Intervention Model Description: Palmar aspect of participants forearms will be randomized to have either a cold compress pack or a room temperature compress pack placed on it. The cold compress pack serves as the trial intervention and the room temperature compress pack serves as the placebo. Each forearm will then be injected with both a 3:1 (experimental ratio) and a 9:1 (standard ratio) mixture of lidocaine with epinephrine:sodium bicarbonate in a randomized order.
Who Masked: Participant
Masking Description: Participants will be blind to the solution ratio of each injection, injector will not be blind to solution to ensure safety.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Left Forearm Injection Sites Cooled, Right Forearm Injection Sites at Room Temperature (Experimental): Palmar aspect of participants left forearm will have a cold compress pack placed on it. The palmar aspect of the right forearm will have a room temperature compress pack placed on it. Each forearm will be injected with 1mL of lidocaine with epinephrine buffered with sodium bicarbonate. Each forearm will be injected once with the experimental ratio (3:1) and once with the standard control ratio (9:1). Injections will be administered in a randomized order.
  Interventions: Other: Cold Compress Pack; Other: Room Temperature Compress Pack; Drug: Lidocaine Epinephrine
- Right Forearm Injection Sites Cooled, Left Forearm Injection Sites at Room Temperature (Experimental): Palmar aspect of participants right forearm will have a cold compress pack placed on it. The palmar aspect of the left forearm will have a room temperature compress pack placed on it. Each forearm will be injected with 1mL of lidocaine with epinephrine buffered with sodium bicarbonate. Each forearm will be injected once with the experimental ratio (3:1) and once with the standard control ratio (9:1). Injections will be administered in a randomized order.
  Interventions: Other: Cold Compress Pack; Other: Room Temperature Compress Pack; Drug: Lidocaine Epinephrine

INTERVENTIONS:
Other: Cold Compress Pack — Palmar aspect of forearm will have a cold compress pack placed on it.
Other: Room Temperature Compress Pack — Palmar aspect of forearm will have a room temperature compress pack placed on it.
Drug: Lidocaine Epinephrine — Lidocaine with epinephrine will be buffered 3:1 with sodium bicarbonate
  Other Names: Lidocaine Epinephrine buffered with Sodium Bicarbonate
Drug: Lidocaine Epinephrine — Lidocaine with epinephrine will be buffered 9:1 with sodium bicarbonate
  Other Names: Lidocaine Epinephrine buffered with Sodium Bicarbonate

SUMMARY:
Participants will have local anesthesia administered to the palmar aspect of both forearms using 4 different injection methods in order to determine which method provides the best results in terms of perceived pain, overall comfort, and participant preference. Injection site cooling and solution buffering using a 3:1 ratio will be compared to the current standard, no injection site cooling and 9:1 solution buffering.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures
* Any gender, aged 21 - 65
* In good general health with no peripheral neuropathy or disorders that may produce peripheral neuropathy such as uncontrolled diabetes mellitus
* Healthy intact skin on the palmar aspect of both left and right forearms
* Fluent in English

Exclusion Criteria:

* Current use of any medication
* Pregnancy
* Known allergic reactions to components of the local anesthetic such as sulfites
* History of vasovagal response to venipuncture or vaccination
* History of trauma to the forearms i.e., bone breaks, burns, deep lacerations
* Decreased sensation to the palmar aspect of either forearm

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Pain from Needle Insertion | 2 Months
  Pain from needle insertion during each injection will be scored on a 0 - 10 scale by participants
Pain from Solution Deposition | 2 Months
  Pain from solution deposition during each injection will be scored on a 0 - 10 scale by participants
Overall Comfort Level During Injection | 2 Months
  Comfort level during each injection will be scored on a 0 - 10 scale by participants

SECONDARY OUTCOMES:
Injection Method Preference | 2 Months
  Participants will select which of the 4 injection methods they preferred

OTHER OUTCOMES:
Buffered Anesthetic Solution pH | 2 Months
  pH of each solution will be measured using a calibrated pH probe

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Bastidas, MD, Principal Investigator — Northwell Health

IPD SHARING:
Plan to Share IPD: No